CLINICAL TRIAL: NCT04990414
Title: Cognitive Behaviour Therapy for Voices and Dissociation: A Case Series
Brief Title: Cognitive Behaviour Therapy for Voices and Dissociation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Filippo Varese, Senior Clinical Lecturer, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: x145-119388
Record Dates: First submitted 2021-06-24; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia; Psychological Trauma; Dissociation; Hallucinations
MeSH Terms: conditions — Schizophrenia; Psychological Trauma; Dissociative Disorders; Hallucinations | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT for voices and dissociation (Experimental): 24 sessions of Cognitive Behavioural Therapy (CBT) over a 6-month period treatment window.
  Interventions: Other: Cognitive Behavioural Therapy

INTERVENTIONS:
Other: Cognitive Behavioural Therapy — Sessions 1-4 were focused on engagement, assessment of presenting problems, identification of treatment goals and normalization/ psychoeducation. Sessions 5- 14, focused on techniques to manage dissociative responses and/or increase perceived controllability of dissociation. Although further work on dissociation and/or trauma was encouraged, the targets for intervention in subsequent sessions (15-22) and the strategies selected depended on individual formulation of clients' difficulties and negotiation with the client. This could include re-appraisals on negative beliefs about dissociative experiences, cognitive and/or behavioural change strategies targeting core appraisals of voices leading to related distress, trauma-related techniques (e.g., imagery techniques,), or consolidation of a developmental/longitudinal psychological formulation of the client's difficulties. The final two sessions focused on plans for relapse prevention and maintenance of gains.

SUMMARY:
Case series design with participants with psychosis with a history of interpersonal trauma/abuse and current distressing auditory verbal hallucinations and dissociative experience. Participants were offered up to 24 therapy sessions over a 6-month intervention window.

DETAILED DESCRIPTION:
Objectives: Previous studies have suggested that dissociation might represent an important mechanism in the maintenance of auditory verbal hallucinations (i.e., voices) in people who have a history of traumatic life experiences. This study investigated whether a cognitive behavioural therapy (CBT) intervention for psychosis augmented with techniques specifically targeting dissociative symptoms could improve both dissociation and auditory hallucination severity in a sample of voice hearers with psychosis and a history of interpersonal trauma (e.g., exposure to sexual, physical, and/or emotional abuse).

Design: Case series.

Methods: A total of 19 service users with psychosis were offered up to 24 therapy sessions over a 6-month intervention window. Participants were assessed four times over a 12-month period using measures of dissociation, psychotic symptoms severity, and additional secondary mental-health and recovery measures.

ELIGIBILITY:
Inclusion Criteria:

1. Be in contact with mental health services.
2. Have an identified care coordinator.
3. Meet ICD-10 criteria for schizophrenia, schizoaffective disorder or delusional disorder or meet entry criteria for an Early Intervention in Psychosis service in order to allow for diagnostic uncertainty in early phases of psychosis.
4. History of voice-hearing for a minimum of six months.
5. Aged 16 and above.
6. Score ≥ 2 (i.e. "Voices occurring at least once a day") on the frequency item of the PSYRATS.
7. Score ≥ 3 (i.e. "Voices are very distressing, although subject could feel worse") on the distress intensity rating of the PSYRATS.
8. Confirmed that they consider AVHs, dissociative experiences, and/or trauma as their main problem or presenting difficulty, and that would like to receive a psychological intervention specifically designed to address these difficulties - this will be assessed using four items integrated in the PSYRATS interview administered as part of the present study, and the self-reported therapy goals generated through the CHOICE short form.
9. Score ≥ 1 on any of the items of the Bref Betrayal Trauma Survey assessing lifetime exposure to interpersonal trauma (i.e. items 3-11).
10. scores suggestive of clinical levels of dissociative symptoms, as indicated by a score > 20 on the Dissociative Experiences Scale, time bound
11. Capacity to provide informed consent.
12. Judged by their clinician to be clinically stable for the preceding 4 weeks

Exclusion Criteria:

1. Any person without capacity to provide written informed consent.
2. If the experience of voices/psychosis is organic in origin (for example, hallucinatory experiences linked to traumatic brain injuries, organic psychoses, or emerging in the context of dementing conditions).
3. Insufficient command of English to complete the research interviews and measures.
4. Intellectual disability, or severe cognitive dysfunction that might preclude the individual's ability to provide informed consent, understand the study procedure and/or fully appreciate the potential consequences of their participation.
5. Primary diagnosis of substance misuse dependency.
6. Where care coordinators identify reasons for why participation might be potentially detrimental.
7. Inpatient/acute care needed.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-11-24 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Change in the Dissociative Experiences Scale - time bound | baseline, at mid-treatment (approximately 3 months after the baseline assessment), at the end of treatment (6 months after baseline), and again at 6 months following the end of treatment
  Change in the frequency of dissociative experiences, assessed via a questionnaire measure assessing presence and frequency of dissociative experiences in the previous month
Change in the Psychotic Symptoms Rating Scale - auditory hallucinations subscale | baseline, at mid-treatment (approximately 3 months after the baseline assessment), at the end of treatment (6 months after baseline), and again at 6 months following the end of treatment
  change in the severity of hallucinatory experiences, assessed via a clinical interview measuring for presence and severity of auditory hallucinations in the previous week

SECONDARY OUTCOMES:
Change in the Psychotic Symptoms Rating Scale - delusions subscale | baseline, at mid-treatment (approximately 3 months after the baseline assessment), at the end of treatment (6 months after baseline), and again at 6 months following the end of treatment
  change in the severity of delusional beliefs, assessed via a clinical interview measuring for presence and severity of delusions in the previous week
Change in the Impact of Events Scale Revised | baseline, at mid-treatment (approximately 3 months after the baseline assessment), at the end of treatment (6 months after baseline), and again at 6 months following the end of treatment
  change in the severity of post-traumatic symptoms, assessed via a questionnaire measuring arousal, hypervigilance, and intrusions in the previous week
Change in the short Depression, Anxiety and Stress Scales | baseline, at mid-treatment (approximately 3 months after the baseline assessment), at the end of treatment (6 months after baseline), and again at 6 months following the end of treatment
  change in the severity of emotional distress, assessed via a questionnaire measuring symptoms of anxiety, depression, and stress in the previous week
Change in the Questionnaire about the Process of Recovery | baseline, at mid-treatment (approximately 3 months after the baseline assessment), at the end of treatment (6 months after baseline), and again at 6 months following the end of treatment
  change in subjective recovery from psychosis, assed via a self-report questionnaire measuring perceived recovery from psychosis-related difficulties
Change in the short-form of the CHoice of Outcome In Cbt for psychosEs (CHOICE) | baseline, at mid-treatment (approximately 3 months after the baseline assessment), at the end of treatment (6 months after baseline), and again at 6 months following the end of treatment
  change in service user-led outcome measure, assessed using a validated questionnaire developed to evaluate outcomes of cognitive behavioural interventions for psychosis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Varese F, Douglas M, Dudley R, Bowe S, Christodoulides T, Common S, Grace T, Lumley V, McCartney L, Pace S, Reeves T, Morrison AP, Turkington D. Targeting dissociation using cognitive behavioural therapy in voice hearers with psychosis and a history of interpersonal trauma: A case series. Psychol Psychother. 2021 Jun;94(2):247-265. doi: 10.1111/papt.12304. Epub 2020 Sep 10. PMID 32914542